CLINICAL TRIAL: NCT02490709
Title: Local Excision of Clinical T3 Mid- or Low-Rectal Adenocarcinoma Showing Major Response(ycT0-1) After Neoadjuvant Chemoradiotherapy: Prospective Multicenter Single-arm Phase II Clinical Trial
Brief Title: Local Excision of Clinical T3 Rectal Adenocarcinoma Showing Major Response(ycT0-1) After Neoadjuvant Chemoradiotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Jae Hwan Oh, Director, Hospital, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-LE
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Rectal Cancer
Keywords: Rectal neoplasms; Colorectal neoplasms; Local excision
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Local excision (Experimental): Local excision for rectal cancer with good response
  Interventions: Procedure: Local excision

INTERVENTIONS:
Procedure: Local excision — Local excision for rectal cancer with good response

SUMMARY:
The purpose of this study is evaluation of the safety and the efficacy of transanal local excision in patients with cT3 rectal cancer which was downstaged into ycT0-1 after neoadjuvant chemoradiotherapy.

DETAILED DESCRIPTION:
This study is a prospective multicenter single-arm phase II clinical trial. Rectal cancer patients with cT3 stage will receive neoadjuvant chemoradiotherapy, and be evaluated the response of the tumor in 6 to 10 weeks after completion of neoadjuvant chemoradiotherapy. For those who have good response (ycT0-1) will underwent transanal local excision under the patients' agree.

ELIGIBILITY:
Inclusion Criteria:

* age: more than 20 years
* biopsy-proven adenocarcinoma of the rectum
* clinical staging, cT3NxM0
* Rectal cancer located 8 cm from the anal verge
* Restaging in 6-10 weeks after completion of neoadjuvant chemoradiotherapy, ycT0-1N0M0
* ECOG performance status 2 or less

Exclusion Criteria:

* Synchronous colon cancer or other malignancy
* Obstructing rectal cancer
* Pregnant or breast-feeding
* Receiving any other study agents
* History of prior colorectal cancer or inflammatory bowel disease
* Hereditary colorectal cancer (FAP, HNPCC)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 1-5 years
  Death or recurrence as an event

SECONDARY OUTCOMES:
Complete response rate | 1-5 years
  The rate of complete response of the tumor after neoadjuvant chemoradiotherapy
Overall survival rate | 1-5 years
  Death as an event

CONTACTS AND LOCATIONS:
Overall Officials: Oh Jae Hwan, MD, PhD, Principal Investigator — National Cancer Center, Republic of Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea